CLINICAL TRIAL: NCT06562452
Title: Evaluating the Effect of Injectable Platelet Rich Fibrin on Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LeNguyenLamCTUMP
Record Dates: First submitted 2024-08-08; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Angle Class I
Keywords: injectable platelet-rich fibrin; canine retraction; orthodontic tooth movement
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: This study was a split-mouth randomized clinical trial was conducted on 31 patients (9 male, 22 females age ranging 14-31 years) who were treated for Class I malocclusion with the extraction of the maxillary first premolar. After the leveling and alignment phase, the canines were retracted with 150gm forces. The i-PRF was prepared from the blood of each patient then injected immediately before canine retraction on the buccal and palatal aspects of the extraction sites. Digital model were obtained at five time points: before tooth extraction (T0) and in the fourth week (T1), eighth week (T2), twelfth week (T3), sixteenth week (T4) from the beginning of distalization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right sides were randomly allocated to treatments with i-PRF (Experimental): The amount of i-PRF was standardized as 2mL and was injected submucosal into the distobuccal and distopalatal side of the canine tooth (1mL for each side) under local anesthesia for pain control.
  Interventions: Diagnostic Test: Injectable platelet rich fbirin
- Left sides were randomly allocated to control sides. (Experimental): The placebo was standardized as 2mL and was injected submucosal into the distobuccal and distopalatal side of the canine tooth (1mL for each side) under local anesthesia for pain control.
  Interventions: Diagnostic Test: Injectable platelet rich fbirin

INTERVENTIONS:
Diagnostic Test: Injectable platelet rich fbirin — fter the leveling and alignment phase, the canines were retracted with 150gm forces. The i-PRF was prepared from the blood of each patient then injected immediately before canine retraction on the buccal and palatal aspects of the extraction sites. Digital model were obtained at five time points: before tooth extraction (T0) and in the fourth week (T1), eighth week (T2), twelfth week (T3), sixteenth week (T4) from the beginning of distalization.

SUMMARY:
Introduction: Prolonged orthodontic treatment can lead to challenges and unfavourable outcomes, including increased risk of caries, root resorption, as well as gingival and periodontal diseases. Acceleration of this step would reduce overall treatment time, improve patient cooperation, and decrease possible negative side effects. The injectable platelet - rich fibrin is second generation holds the advantages of easier preparations and longer effects that is obtained through low-speed centrifugation. The potential benefits of PRF have been widely investigated in regenerative dentistry and oral surgery such as tooth movement, implantology, oral pathology and periodontal therapy.

Objective: Our study aims to investigate the effectiveness of i PRF in accelerating maxillary canine retraction Subjects and method: This study was a split-mouth randomized clinical trial was conducted on 31 patients (9 male, 22 females age ranging 14-31 years) who were treated for Class I malocclusion with the extraction of the maxillary first premolar. After the leveling and alignment phase, the canines were retracted with 150gm forces. The i-PRF was prepared from the blood of each patient then injected immediately before canine retraction on the buccal and palatal aspects of the extraction sites. Digital model were obtained at five time points: before tooth extraction (T0) and in the fourth week (T1), eighth week (T2), twelfth week (T3), sixteenth week (T4) from the beginning of distalization.

DETAILED DESCRIPTION:
One of the main goals of orthodontic treatment is the reduction of treatment time through faster tooth movement, acceleration of canine retraction and space closure would reduce overall treatment time. Tooth movement is essentially a biological response to a physical stimulus, speeding up this response should avoid the occurrence of common iatrogenic effects such as white spot lesions, caries, root resorption and periodontal problems 1. Therefore, attempts to accelerate tooth movement and reduce treatment duration are of great significance to both orthodontists and patients. Thus, various invasive and non-invasive modalities have been attempted to reduce the duration of orthodontic treatment by accelerating tooth movement such as: surgical, vibration, pharmacological agents, low-level laser therapy or other procedures 2,3,4,5. However, none of these procedures have yet become a gold standard method. Platelet-based preparations from the patient's blood provide a safe alternative to commercially available bioactive materials. Platelet-rich fibrin (PRF) is the second generation, holds the advantages of easier preparations and longer effects 6-11. The injectable platelet-rich fibrin (i-PRF) was developed as an advanced product of PRF by altering the centrifugation protocol by lowering the centrifugation speed and force to 700 rotations per minute within 3 minutes. has many advantages over the conventional form such as higher rates of leukocyte, regenerative cells and growth factors. The potential benefits of PRF have been widely investigated in regenerative dentistry and oral surgery such as tooth movement, implantology, oral pathology and periodontal therapy 12,13,14. Wang et al. reported that i-PRF affected osteoblastic behavior remarkably by influencing its migration, proliferation, and differentiation. This promotes cellular activity and accelerates bone turnover and healing 11.

The purpose of this study was to investigate the efficiency of i-PRF in accelerating tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* Participants (age>12 years old) with Class I malocclusion requiring extraction of maxillary first premolar
* No previous orthodontic treatment
* Absence of systemic diseases and dentofacial anomalies
* Participant agreed to participate in the study

Exclusion criteria:

* Participants with periodontal diseases, craniofacial syndromes such as cleft lip or palate, systemic diseases related to bone metabolism
* Taking anticoagulants or medication that interferes with orthodontic tooth movement for example, heparin, warfarin, NSAIDs, cyclosporine, glucocorticoids, medroxyprogesterone acetate, thyroid hormones,

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
The purpose of this study was to investigate the efficiency of i-PRF in accelerating tooth movement. | Our study aims to investigate the effectiveness of i PRF in accelerating maxilary canine retraction at 5 time points (5 months): before tooth extraction (T0) and in the fourth week (T1), eighth week (T2), twelfth week (T3), sixteenth week (T4)
  Digital models were scanned using the iTero scanner (Align Technology, Inc, USA) assessed by Medit Link software at 5 time points (5 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

REFERENCES:
- [Result] Erdur EA, Karakasli K, Oncu E, Ozturk B, Hakki S. Effect of injectable platelet-rich fibrin (i-PRF) on the rate of tooth movement. Angle Orthod. 2021 May 1;91(3):285-292. doi: 10.2319/060320-508.1. PMID 33459765